CLINICAL TRIAL: NCT01479010
Title: Pilot Study of the Safety and Efficacy of Anakinra (Recombinant Human Interleukin-1 Receptor Antagonist) in Pulmonary Hypertension
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: recruitment issues, critical investigators left institution
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM13729
Record Dates: First submitted 2011-11-07; First posted 2011-11-24 (Estimated); Results first posted 2015-06-08 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-10

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Anakinra (Experimental)
  Interventions: Drug: Anakinra 100 mg subcutaneously daily

INTERVENTIONS:
Drug: Anakinra 100 mg subcutaneously daily — Anakinra 100 mg subcutaneously daily

SUMMARY:
This is an open-label non-randomized, pilot study to evaluate the effect of Interleukin-1 blockade on exercise capacity in patients with pulmonary hypertension. Subjects will undergo cardiopulmonary exercise testing at baseline, and after 4 weeks treatment with Anakinra (recombinant human Interleukin-1 receptor antagonist.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Diagnosis of PAH (from prior right heart catheterization), with functional class III symptoms of right ventricle failure despite optimal PAH therapy
* Mean pulmonary artery pressure >25 mmHg
* Pulmonary capillary wedge pressure <15 mmHg
* Pulmonary vascular resistance >3 wood units

Exclusion Criteria:

* PAH due to connective tissue disease (including scleroderma), interstitial lung disease (total lung capacity <65% predicted value), or cirrhosis (portopulmonary hypertension)
* Angina or electrocardiograph (ECG) changes that limit maximum exertion during cardiopulmonary exercise testing or baseline ECG changes that limit the ability to detect ischemia (i.e. left bundle-branch block).
* Recent (<14 days) use of anti-inflammatory drugs (not including NSAIDs), chronic inflammatory disorder (including but not limited to rheumatoid arthritis, systemic lupus erythematosus), malignancy, active infection, or any comorbidity limiting survival or ability to complete the study
* Severe kidney dysfunction (eGFR <30 mL/min)
* Thrombocytopenia (<50,000/mm3), or neutropenia (absolute neutrophil count <1,500/mm3)
* Refusal by a woman of childbearing potential (not post-menopausal or surgically sterile) to use a medically acceptable form of birth control (including, but not limited to, a diaphragm, an intrauterine device (IUD), progesterone implants or injections, oral contraceptives, the double-barrier method, or a condom) throughout the duration of the study
* History of hypersensitivity to anakinra or E. coli products
* Latex or rubber allergy
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-11; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Van Tassell, Pharm D., Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Anakinra
Started | 2
Completed | 1
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: Due to the small number of participants, results are not included to protect the privacy of individual participants.
Arm/Group | Anakinra
Number analyzed (Participants) | 0
Age, Continuous [unit: years]
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Median Interval Change From Baseline in Peak VO2
Description: Peak VO2 will be measured during a standardized cardiopulmonary exercise test in which patients exercise on a treadmill while breathing through a mask.
Time Frame: 28 days
Population: Due to the small number of participants, results are not included to protect the privacy of individual participants.
Arm/Group | Anakinra
Number analyzed (Participants) | 0

2. Primary Outcome: Median Interval Change From Baseline in the Minute Ventilation and Carbon Dioxide Production (VE/VCO2 Slope)
Description: VE/VCO2 slope will be measured during a standardized cardiopulmonary exercise test in which patients exercise on a treadmill while breathing through a mask.
Time Frame: 28 days
Population: Due to the small number of participants, results are not included to protect the privacy of individual participants.
Arm/Group | Anakinra
Number analyzed (Participants) | 0

3. Secondary Outcome: Interval Change From Baseline in Biomarkers (High-sensitivity C-reactive Protein, Whole Blood Assay, Brain Natriuretic Peptide)
Time Frame: 28 days
Population: Due to the small number of participants, results are not included to protect the privacy of individual participants.
Arm/Group | Anakinra
Number analyzed (Participants) | 0

4. Secondary Outcome: Interval Change From Baseline in Heart Failure Symptoms as Measured by Duke Activity Status Index (DASI)
Time Frame: 28 days
Population: Due to the small number of participants, results are not included to protect the privacy of individual participants.
Arm/Group | Anakinra
Number analyzed (Participants) | 0

5. Secondary Outcome: Correlation Between Interval Changes in Biomarkers, Peak VO2, and VE/VCO2
Time Frame: 28 days
Population: Due to the small number of participants, results are not included to protect the privacy of individual participants.
Arm/Group | Anakinra
Number analyzed (Participants) | 0

6. Secondary Outcome: Rate of Adverse Events and Hospitalizations
Time Frame: 28 days
Population: Due to the small number of participants, results are not included to protect the privacy of individual participants.
Arm/Group | Anakinra
Number analyzed (Participants) | 0

7. Secondary Outcome: Total Exercise Time
Time Frame: 28 days
Population: Due to the small number of participants, results are not included to protect the privacy of individual participants.
Arm/Group | Anakinra
Number analyzed (Participants) | 0

8. Secondary Outcome: Oxygen Uptake Efficiency Slope
Time Frame: 28 days
Population: Due to the small number of participants, results are not included to protect the privacy of individual participants.
Arm/Group | Anakinra
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Anakinra
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 1/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anakinra (N=2)
Injection site reaction (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes